CLINICAL TRIAL: NCT03762070
Title: Evaluation of a Diagnostic Device, CL Detect™ Rapid Test, for the Diagnosis of Cutaneous Leishmaniasis in Peru
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Max Grogl, Scientific Director, Naval Medical Research Center
Other Study IDs: LRDD-PERU-02
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: CL Detect™ Rapid Test — Observational study of a FDA cleared device, the CL Detect™ Rapid Test.

SUMMARY:
Determine the sensitivity and specificity of the FDA-cleared CL Detect™ Rapid Test in Peru, using a test procedure that was modified from that described in the device instructions to optimize these parameters for the detection of Leishmania species identified in Peru.

DETAILED DESCRIPTION:
Observational study of a FDA cleared device, the CL Detect™ Rapid Test. Data for the 510(K) was supported by a sensitivity study conducted in Tunisia, Old world Leishamania major and a specificity study conducted in the United Sates. Sensitivity and specificity data collected recently in Peru (2014-2015), by the Instituto de Medicina Tropical Alexander von Humbolt, supports the idea that the sensitivity of the CL Detect™ Rapid Test can be drastically increased for New World Leishmania species. The study is a single trial, with two clinical sites, NAMRU-6, Puerto Maldonado and the Alexander von Humboldt Tropical Medicine Institute in Lima. The objective of the study is to determine the sensitivity and specificity of the FDA-cleared CL Detect™ Rapid Test, using an optimized test procedure determined from a pilot study conducted in Peru. Two modifications to the test procedure (marketed device instructions) are included in this study: 1) increase in extraction time in lysis buffer from 5 to 10 minutes to 20 to 30 minutes and 2) a 20 μl increase in the volume of the sample to add to the test strip, from 20 μl to 40 μl. The gold standard for Leishmania diagnosis, which is microscopic identification of amastigotes in stained lesion sample, will be used as a control.

Participants will be patients who present for medical consultation due to a suspected CL lesion. After obtaining informed consent and screening the participant for eligibility, we will collect and test at most 4 samples from the index lesion in the following order:

1. one sample obtained with a dental broach for use with the CL Detect™ Rapid Test;
2. one sample obtained by scraping for microscopic identification of amastigotes; and
3. one sample obtained by scraping for Leishmania speciation by PCR; and
4. when possible, (depending on the size of the lesion), one sample from a different site of the same lesion, obtained by scraping for use with the CL Detect™ Rapid Test. PCR analysis will be performed by NAMRU-6 for possible exploratory analyses including species identification. If the etiologies of the lesions that are negative for Leishmania are known, they will be reported. Participants with a positive diagnosis of leishmaniasis by microscopy or other methods will be referred for standard of care treatment in Peru by the attending physician of the Peruvian Ministry of Health. Treatment is not part of this study. If a participant's lesions are negative for Leishmania, standard of care follow-up testing will be performed, either at the study site, or (when indicated) in another hospital.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and generally healthy.
* Able to provide written informed consent.
* Index lesion present that is suspicious for CL, as defined by the following criteria for an index lesion:

  1. less than 2 months in age
  2. primarily ulcerative, i.e. not purely verrucous or nodular
  3. no clear clinical evidence of cellulitis
  4. location suitable for collecting samples by dental broach and scraping.
* Capable of understanding and complying with the protocol, in the opinion of the evaluator

Exclusion Criteria:

* Received treatment for leishmaniasis within the last 2 months prior to evaluation.
* In the opinion of the investigator, evidence of manipulation of the lesion.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of male and female participants, ages 18 years and older, with a clinically suspected CL lesion. It is estimated that up to 200 participants may need to be consented, screened, and tested in order to obtain 100 participants/samples who are positive by microscopy for Leishmania, using minimally modified (from the device instructional insert) test conditions determined to be optimal in a pilot study. If a higher percentage of participants are negative by microscopy than is estimated, then the total sample size will be increased to obtain a total of 100 participants positive by microscopy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The performance (sensitivity and specificity) of the CL Detect™ Rapid Test | 1 day
  Sensitivity and specificity of CL Detect™ Rapid Test will be determined by comparing with the gold standard, microscopy of stained lesion samples for identification of Leishmania amastigotes. The following definitions apply to the calculation of assay sensitivity and specificity: 1. True positive: Positive by both the CL Detect™ Rapid Test and the reference method. 2. False positive: Positive by the CL Detect™ Rapid Test but negative for the reference method. 3. True negative: Negative by both the CL Detect™ Rapid Test and the reference method. 4. False negative: Negative by the CL Detect™ Rapid Test but positive for the reference method.

SECONDARY OUTCOMES:
Determine the sensitivity and specificity of the FDA-cleared CL Detect™ Rapid Test when scraping is used to obtain tissue samples. | 1 day
  Determine the sensitivity and specificity of the FDA-cleared CL Detect™ Rapid Test when scraping is used to obtain tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Max Grogl, Ph.D., Principal Investigator — Scientific Director
Locations (2):
- Peru (2):
  - Universidad Peruana Cayetano Heredia (UPCH), Lima
  - U.S. Naval Medical Research Center Unit No. 6 (NAMRU-6), Puerto Maldonado

REFERENCES:
- [Derived] Grogl M, Joya CA, Saenz M, Quispe A, Rosales LA, Santos RDP, De Los Santos MB, Donovan N, Ransom JH, Ramos A, Llanos Cuentas E. Evaluation of a diagnostic device, CL Detect rapid test for the diagnosis of new world cutaneous leishmaniasis in Peru. PLoS Negl Trop Dis. 2023 Mar 13;17(3):e0011054. doi: 10.1371/journal.pntd.0011054. eCollection 2023 Mar. PMID 36913433